CLINICAL TRIAL: NCT01981434
Title: Technology Based Obesity Prevention Project (TeBOPP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valleywise Health (Other)
Collaborators: Arizona State University (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013-132
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Obesity in Children
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video game based obesity education (Active Comparator): This is the intervention group. They will be given the opportunity to play an interactive educational video game for teaching health and nutrition.
  Interventions: Other: Video game based obesity education
- No intervention (No Intervention): This is the control group that will receive only printed information about health and nutrition and will not be given the opportunity to play the educational video game.

INTERVENTIONS:
Other: Video game based obesity education — The intervention will be in the form of a videogame in which both parent and their children will participate. The game incorporates lessons from research on avatars (e.g., the Proteus Effect), and game dynamics to explore ways to increase healthy eating and exercise.
  Arms: Video game based obesity education

SUMMARY:
Technology-Based Obesity Prevention Project (TeBOPP) is a bilingual (English/Spanish) family-based educational intervention that will use a novel videogame format to educate underserved inner city Latino children and adolescent patients and their parents about healthy diet and exercise. To the best of our knowledge this is the first family focused obesity prevention educational intervention using a gaming scenario where both parents and children/teens (8-15 years) participate simultaneously. The goals are to improve parent-child (teen) knowledge regarding healthy food habits and create a change in attitude towards healthy eating and exercise.

Hypothesis: We hypothesize that game-based avatars (i.e., a graphical representation of an individual within a virtual space) can create change in knowledge and attitude towards healthy eating and exercise.

DETAILED DESCRIPTION:
Childhood obesity has reached epidemic proportions in recent years and has become the number one challenge among child healthcare providers in the United States. Unhealthy dietary habits and lack of physical activity are among the key factors attributed to increase in overweight and obesity rates among children and adolescents. Obesity is associated with a much higher risk for chronic medical conditions and increasingly diseases among the old like diabetes is becoming commonplace among the young. This growing epidemic may prove to have a tremendous societal impact and may prove to be a colossal economic and health burden in the future if it is not confronted aggressively at this stage. Unfortunately the obesity epidemic has affected the minority and socio economically deprived population in a disproportionate manner. Inner city Latino children and adolescents are being increasingly affected and targeted intervention for this population group is of paramount importance.

In this project, we intend to study the role of an immersive video game technology using simulated game-based avatars to educate parents and children simultaneously about the importance of healthy diet and exercise, assess knowledge gained and retention and their change in attitudes towards adoption of a healthier lifestyle.

Such an innovative educational model deployed using a bilingual (English/Spanish) videogame format which is a natural draw for this age group will likely capture their attention and be successful in conveying the intended message encouraging adoption of healthy diet and exercise. By encouraging parental participation, knowledge gained is expected to be shared and encourage parent-child discussion thereby fostering a team effort to combat obesity and promote a healthy lifestyle in the family as a whole.

The intervention will be specifically tailored to its target population for better acceptance. Our patient population primarily comprises of Mexican-American children and families and issues relating over weight and obesity are most problematic in this population group. A Needs Assessment Survey will be conducted at the start of the project and socio-cultural attributes impacting diet and exercise habits will be assessed. This information will be used to address these specific issues in the game design. If this culturally and linguistically responsive obesity prevention educational intervention for Latino children and families proves a success, future research will focus on making the application easily downloadable on to a mobile internet device for dissemination to a much larger audience. Since the proposed intervention is based on the concepts of cognitive behavior therapy, opportunities for repeat play is likely to reinforce knowledge gain and encourage a positive health behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Latino ethnicity, 8 to 15 years of age who register in the pediatric ED and patients who visit the three FLCs and are accompanied by a parent/guardian who is 18 years or older and able to communicate in English or Spanish
* A patient must receive an Emergency Severity Index (ESI) Version 3 score of 4/5 indicating non-urgent status for recruitment in the pediatric ED.

Exclusion Criteria:

* Medically unstable patients (in the pediatric ED), patients with ESI score of 1-3 (life threatening medical/surgical condition).
* Incarcerated patients or patients from juvenile detention facilities.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2016-07-26 (Actual)

PRIMARY OUTCOMES:
Improvement in knowledge regarding a healthy diet and nutrition among parents/children using a video game based educational intervention | 18 months
  Nutrition knowledge measured by change in each subject's scores on pre and post tests developed by the investigator especially for this study.

SECONDARY OUTCOMES:
Improvement in parent/child communication and intent to adopt a healthier lifestyle using a video game based educational intervention | 18 months
  Improvement in communication levels were obtained with pre and post satisfaction surveys

OTHER OUTCOMES:
Game usage time up to completion. | 18 months
  Game usage was tracked throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Coonrod, MD, Principal Investigator — District Medical Group
Locations (1):
- Maricopa Integrated Health System, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No